CLINICAL TRIAL: NCT01669031
Title: Effect of Exposure to Computer Simulated Visual Field Testing on Variability and Reliability of Test Results: A Randomized Controlled Trial
Brief Title: Randomized Controlled Trial on Visual Field Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oftalmologia Hospital Sotero del Rio (Other)
Responsible Party: Principal Investigator, Eugenio A. Maul, Investigator, Oftalmologia Hospital Sotero del Rio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Oftalmo_Glaucoma_002
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Glaucoma
Keywords: automated perimetry; visual fields; reliability; vision tests/standards; randomized controlled trial; false positive reactions; false negative reactions; fixation, ocular; mean deviation; variability; program; software; glaucoma/diagnosis; visual field tests/methods; aged; humans; female; male; prospective studies; reproducibility of results
MeSH Terms: conditions — Glaucoma; Disease

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): No practice tests are performed in this arm
- Practice Program (Experimental): At the 3 study visits exposed to a training session (simulated visual field test on a computer).
  Visit 1 they get 2 simulated tests tests per eye. At visits 2 and 3 they get 1 simulated test per eye. Each simulated test takes 3-15 minutes
  Interventions: Other: Practice program

INTERVENTIONS:
Other: Practice program — Each practice session (simulated visual field test on computer) takes 3-15 minutes
  Other Names: Computer Simulated practice Visual Field Test
  Arms: Practice Program

SUMMARY:
Unreliability and visual field variability is a known problem with automated perimetry in both developing and developed country settings. This study will look at the effects of a computer program that allows new patients to practice the visual field exam before taking the actual exam. Our hypothesis is that the intervention group will have less variability as measured by mean deviation between exams and greater reliability as measured by the standard unreliability indexes of false positive rate, false negative rate, and fixation losses.

DETAILED DESCRIPTION:
3 study visits. Visit 1: Baseline visit for consent, getting baseline data and finally randomizing the patient. Those randomized to intervention get their first session of simulated visual field (2 per eye) on a regular computer for training purposes.

Visit 2: 1 to 2 days after baseline. The intervention group gets 1 practice test per eye. Then both groups get a regular automated visual field Visit 3: 1 to 2 weeks after baseline. The intervention group gets 1 practice test per eye. Then both groups get a regular automated visual field.

Study Ends, patient gets seen by the patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or greater
* Referred to the glaucoma clinic for examination due to suspected glaucoma or glaucoma diagnosis
* No more than 1 automated visual field test within the last 4 years

Exclusion Criteria:

* patients who cannot remain seated for 10 minutes
* patients with neck problems that prevent them from using the field analyzer properly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
The absolute value of the difference in mean deviation of the first and second visual field exam | Visual field exams obtained 1 to 2 weeks apart

SECONDARY OUTCOMES:
Difference in the absolute number of altered points in the visual field with a total deviation below the 0.5 percentile | Visual field exams obtained 1 to 2 weeks apart
Difference in the percentage of false positives, false negatives, and fixation losses at the first and second exam between control and intervention group | Visual field exams obtained 1 to 2 weeks apart
Difference in the time required to complete the first and second exam | Visual field exams obtained 1 to 2 weeks apart
Difference in the proportion of unreliable visual fields at the first and second exam between control and intervention groups | Visual field exams obtained 1 to 2 weeks apart

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sótero del Río, Santiago, Puente Alto, Chile